CLINICAL TRIAL: NCT00312065
Title: Servocontrolled Radiant Warmers and the Role of Thermistor Probe Reflective Shields in Neonates
Brief Title: Study of the Need for Temperature Probe Covers for Newborn Babies on Radiant Warmers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Alan de Klerk, Associate Director of Neonatology, Maimonides Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #03/10/VA03
Record Dates: First submitted 2006-04-05; First posted 2006-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Impaired Thermoregulation
Keywords: servocontrolled; radiant warmer; thermistor; heat shield

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental): Once stabilized, a trimmed reflective shield to cover only the probe itself will be placed over the thermistor probe. Changes in measured skin temperature and warmer power output will be recorded non-invasively, as well as the time taken to reestablish baseline status. A full-sized reflective shield will then be placed over the thermistor probe and the same observations recorded, then repeated 15 minutes later. At the time of a subsequent routine change in thermistor position, the same procedure will be followed, but omitting the intermediate step of using the smaller trimmed shield. Continuous core temperatures will be monitored via a short rectal probe during the study periods.
  Interventions: Device: Application of reflective heat shield to thermistor probe

INTERVENTIONS:
Device: Application of reflective heat shield to thermistor probe

SUMMARY:
The purpose of this study is to examine the need for reflective heat shield covers over the temperature probes applied to the skin of newborn babies who are being nursed under a radiant warmer.

DETAILED DESCRIPTION:
Servocontrolled radiant warmers are widely used for infants' temperature maintenance. Covering the attached skin temperature (or thermistor) probe with a reflective shield may prevent inadvertent warming of the probe by the radiant heat source. However the shield itself might cause falsely elevated or lowered measured skin temperatures, and the use of such shields, while widespread, is not universal nor standard of care. This study aims to document the effects of a reflective shield on the measured skin temperatures of neonates nursed under radiant warmers.

Stable newborn infants in the Maimonides NICU who are being nursed under a radiant warmer will be studied. As part of routine care, the thermistor probe will be applied and the desired servocontrolled skin temperature set. Once stabilized, a trimmed reflective shield to cover only the probe itself will be placed over the thermistor probe. Changes in measured skin temperature and warmer power output will be recorded non-invasively, as well as the time taken to reestablish baseline status. A full-sized reflective shield will then be placed over the thermistor probe and the same observations recorded, then repeated 15 minutes later. At the time of a subsequent routine change in thermistor position, the same procedure will be followed, but omitting the intermediate step of using the smaller trimmed shield. Continuous core temperatures will be monitored via a short rectal probe during the study periods.

The effect of the use of the different size temperature probes will be examined by analyzing the effect on measured skin temperature.

ELIGIBILITY:
Inclusion Criteria:

* Stable newborn infants greater than 1000g birth weight
* On room air or on CPAP in 21% oxygen
* Being nursed under radiant warmer

Exclusion Criteria:

* Major congenital anomalies
* Significant dermatological pathology or abnormalities
* Documented or suspected sepsis

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2003-10; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The effect of the use of the reflective heat shield on the measured skin temperature of the baby

SECONDARY OUTCOMES:
The effect of the use of the reflective heat shield on the measured rectal temperature of the baby
The effect of the use of the reflective heat shield on the measured power output of the radiant warmer

CONTACTS AND LOCATIONS:
Overall Officials: Alan M de Klerk, MBChB, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States